CLINICAL TRIAL: NCT01228136
Title: Use of Tranexamic Acid for Bleeding Reduction in Adenotonsillectomy in Children
Brief Title: Tranexamic Acid and Pediatric Adenotonsillectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Irmandade Santa Casa de Misericórdia de Porto Alegre (Other)
Responsible Party: Marília Ribeiro Brum, Irmandade Santa Casa de Misericórdia de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ISCMPA02
Record Dates: First submitted 2010-10-22; First posted 2010-10-26 (Estimated); Last update posted 2010-12-22 (Estimated); Status verified 2010-10

CONDITIONS: Tonsillectomy; Adenoidectomy; Tranexamic Acid
Keywords: Adenotonsillectomy; Tranexamic acid; Blood loss; Postoperative hemorrhage
MeSH Terms: conditions — Hemorrhage; Postoperative Hemorrhage | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tranexamic acid (Active Comparator)
  Interventions: Drug: Tranexamic Acid
- Placebo (Placebo Comparator)
  Interventions: Other: normal saline solution

INTERVENTIONS:
Drug: Tranexamic Acid — 10mg/Kg, IV (in the vein), first dose 30 minutes before surgery, second dose 8 hours after first dose, third dose 8 hours after second dose
  Other Names: Transamin; Hemoblock
  Arms: Tranexamic acid
Other: normal saline solution — normal saline solution in the same volume calculated as treatment (tranexamic acid 250mg/mL, 10mg/Kg), IV (in the vein) first dose 30 minutes before surgery, second dose 8 hours after first dose, third dose 8 hours after second dose
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if the use of tranexamic acid prior adenotonsillectomy in children can reduce surgical and postoperative bleeding.

DETAILED DESCRIPTION:
Tonsillectomy with or without adenoidectomy is the most common major surgical procedure performed in children. Although it's a relatively simple procedure, may present complications as hemorrhage and death. The mortality associated to the surgery range between 1/1.000 and 1/27.000 in the literature, with approximately 30% due to hemorrhage.

Tranexamic acid is an antifibrinolytic hemostatic indicated to control bleeding in cases of hyperfibrinolysis or defective hemostasis diseases. It's major indications are prostatic surgery and menorrhagia.

ELIGIBILITY:
Inclusion Criteria:

* children with 4 to 12 years
* adenotonsillar hypertrophy
* indication of adenotonsillectomy

Exclusion Criteria:

* patients with blood dyscrasia
* patients with history of bleeding of difficult control or spontaneous hematoma
* patients with coagulation tests altered
* patients with evidence of hematopoietic, cardiovascular, hepatic, renal, neurologic, psychiatric or auto immune disease

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 95 (Actual)
Dates: Start 2010-01; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
volume of intraoperative bleeding | one day
  intraoperative bleeding (in mL of aspirated blood) measured at the end of the surgical procedure

SECONDARY OUTCOMES:
incidence of postoperative bleeding | ten days
  incidence of oral bleeding at the ten days after surgery, evaluated by a patient's diary and postoperative medical evaluations

CONTACTS AND LOCATIONS:
Overall Officials: Marília R Brum, MD, Principal Investigator — Irmandade Santa Casa de Misericórdia de Porto Alegre; José Faibes Lubianca Neto, MD, Study Director — Irmandade Santa Casa de Misericórdia de Porto Alegre
Locations (1):
- Hospital da Criança Santo Antônio, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Brum MR, Miura MS, Castro SF, Machado GM, Lima LH, Lubianca Neto JF. Tranexamic acid in adenotonsillectomy in children: a double-blind randomized clinical trial. Int J Pediatr Otorhinolaryngol. 2012 Oct;76(10):1401-5. doi: 10.1016/j.ijporl.2012.04.028. Epub 2012 Jun 16. PMID 22704676